CLINICAL TRIAL: NCT05399303
Title: Pain Evaluation After Single Visit Nonsurgical Retreatment Using a Bio Ceramic Sealer
Brief Title: Bioceramics Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Ghobashy, associate professor, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: END 10 231
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Endodontically Treated Teeth; Post Operative Pain
Keywords: bio-ceramic postoperative pain sealer
MeSH Terms: conditions — Tooth, Nonvital; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioceramic sealer obturation (Experimental)
  Interventions: Procedure: obturation
- resin sealer (Experimental)
  Interventions: Procedure: obturation

INTERVENTIONS:
Procedure: obturation — obturation using different types of sealers

SUMMARY:
Postoperative pain in endodontic retreatment cases presents a challenge to any endodontist. Tricalcium silicate materials as mineral trioxide aggregate (MTA) and bioceramics have shown favorable periapical tissue reactions and healing when used as part of the root canal filling material. This study was conducted to compare the difference in the postoperative pain when resin cements are used versus bioceramic cements in the obturation of root canals.

DETAILED DESCRIPTION:
The Faculty of Dentistry Ain Shams University's Research Ethics Committee reviewed the current proposal for ethical approval. One hundred patients with permanent molar teeth requiring endodontic non-surgical retreatment were treated in this study. Teeth with fractured instruments were excluded. Patient ages ranged from twenty to fifty years, both men and women were treated in the current study. Infants, children, people unable to take decisions, university students, orphans, mentally or physically disabled patients were excluded from the current study.

Preoperative assessment of the degree of the patient's pain was done using the visual analog scale. Fifty teeth were obturated with gutta percha using the epoxy resin-based sealer (AH Plus) as the control group, and in the other fifty bioceramic based cement (Endosequence) was used. All teeth were prepared by the protaper next rotary files (Dentsply Sirona) under copious irrigation with 30ml of 2.6 % sodium hypochlorite throughout the procedure. Ethylamine diamine tetracetic acid (EDTA) 17% was used to remove the smear layer before the obturation commenced. Obturation was done using the cold lateral compaction technique in the resin group and single cone technique in the bioceramic group. Postoperative pain assessment was done for each patient after six hours, twenty-four hours, four days and one week.

ELIGIBILITY:
Inclusion Criteria:

* • Mandibular molars with fully formed roots that need retreatment.

  * Age range 20 - 50 years.
  * Teeth having a baseline periapical lesion (PAI score ≥2) in the affected root.

Exclusion Criteria:

* • Patients with separated files that need to be retrieved or bypassed.

  * Pregnant females.
  * Patients suffering from a systemic disease.
  * Teeth with lesions connected to adjacent teeth.
  * Teeth with root fractures or perforations.
  * Teeth with lesions communicating with the alveolar crest.
  * Patients with generalized chronic periodontitis or teeth that need periodontal surgery prior to coronal restorations due to marginal deficiency
  * Teeth with damaged or resorbed peri- apex
  * Teeth that were treated with a fiber post and teeth with canal curvature more than 30 degrees.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | one week
  Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Locations (1):
- MIU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Data other than personal data will be shared

REFERENCES:
- [Background] Yoldas O, Topuz A, Isci AS, Oztunc H. Postoperative pain after endodontic retreatment: single- versus two-visit treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Oct;98(4):483-7. doi: 10.1016/j.tripleo.2004.03.009. PMID 15472665
- [Background] Comparin D, Moreira EJL, Souza EM, De-Deus G, Arias A, Silva EJNL. Postoperative Pain after Endodontic Retreatment Using Rotary or Reciprocating Instruments: A Randomized Clinical Trial. J Endod. 2017 Jul;43(7):1084-1088. doi: 10.1016/j.joen.2017.02.010. Epub 2017 May 3. PMID 28477995
- [Background] Seltzer S, Naidorf IJ. Flare-ups in endodontics: I. Etiological factors. 1985. J Endod. 2004 Jul;30(7):476-81; discussion 475. doi: 10.1097/00004770-200407000-00005. PMID 15220641
- [Background] Trope M. Flare-up rate of single-visit endodontics. Int Endod J. 1991 Jan;24(1):24-6. doi: 10.1111/j.1365-2591.1991.tb00866.x. PMID 1917085
- [Background] Mattscheck DJ, Law AS, Noblett WC. Retreatment versus initial root canal treatment: factors affecting posttreatment pain. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Sep;92(3):321-4. doi: 10.1067/moe.2001.115135. PMID 11552152
- [Background] Atav Ates A, Dumani A, Yoldas O, Unal I. Post-obturation pain following the use of carrier-based system with AH Plus or iRoot SP sealers: a randomized controlled clinical trial. Clin Oral Investig. 2019 Jul;23(7):3053-3061. doi: 10.1007/s00784-018-2721-6. Epub 2018 Nov 5. PMID 30397735
- [Background] Graunaite I, Skucaite N, Lodiene G, Agentiene I, Machiulskiene V. Effect of Resin-based and Bioceramic Root Canal Sealers on Postoperative Pain: A Split-mouth Randomized Controlled Trial. J Endod. 2018 May;44(5):689-693. doi: 10.1016/j.joen.2018.02.010. Epub 2018 Mar 20. PMID 29571915
- [Background] Drumond JPSC, Maeda W, Nascimento WM, Campos DL, Prado MC, de-Jesus-Soares A, Frozoni M. Comparison of Postobturation Pain Experience after Apical Extrusion of Calcium Silicate- and Resin-Based Root Canal Sealers. J Endod. 2021 Aug;47(8):1278-1284. doi: 10.1016/j.joen.2021.05.008. Epub 2021 May 29. PMID 34058249
- [Background] Materials used for root canal obturation: technical, biological and clinical testingORSTAVIK DEndodontic Topics (2005) 12(1)
- [Background] DiRenzo A, Gresla T, Johnson BR, Rogers M, Tucker D, BeGole EA. Postoperative pain after 1- and 2-visit root canal therapy. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 May;93(5):605-10. doi: 10.1067/moe.2002.121900. PMID 12075212
- [Background] Toia CC, Khoury RD, Corazza BJM, Orozco EIF, Valera MC. Effectiveness of 1-Visit and 2-Visit Endodontic Retreatment of Teeth with Persistent/Secondary Endodontic Infection: A Randomized Clinical Trial with 18 Months of Follow-up. J Endod. 2022 Jan;48(1):4-14. doi: 10.1016/j.joen.2021.09.004. Epub 2021 Sep 20. PMID 34555421